CLINICAL TRIAL: NCT06332404
Title: Hypoglossal Nerve Stimulation (HNS) Therapy in Patients With Obstructive Sleep Apnea (OSA): Belgian Registry
Brief Title: Hypoglossal Nerve Stimulation Therapy in Patients With Obstructive Sleep Apnea: Belgian Registry
Acronym: B-HNS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: B3002024000047
Record Dates: First submitted 2024-03-13; First posted 2024-03-27 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea; Apnea
Keywords: hypoglossal nerve stimulation; registry; routine clinical care
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Obstructive sleep apnea (OSA) patients treated with hypoglossal nerve stimulation (HNS) therapy: OSA patients treated with HNS therapy will be asked to participate in the registry.
  Interventions: Device: Hypoglossal nerve stimulation Inspire system (Inspire Medical Systems Inc., USA)

INTERVENTIONS:
Device: Hypoglossal nerve stimulation Inspire system (Inspire Medical Systems Inc., USA) — Hypoglossal nerve stimulation therapy
  Other Names: Inspire system (Inspire Medical Systems Inc., USA); Inspire device; HNS therapy

SUMMARY:
Hypoglossal nerve stimulation (HNS) therapy (Inspire system) is intended for the treatment of patients with moderate to severe obstructive sleep apnea (OSA) who cannot be effectively treated with the first-line treatment options. Recently, the request for reimbursement of the Inspire system in Belgium was approved.

The aim is to create a multi-center registry of OSA patients that are treated with HNS (Inspire system) within routine clinical care in Belgium.

DETAILED DESCRIPTION:
Patients that are implanted with the Inspire system in Belgium will be invited to participate in the registry. Data will be collected from different routine clinical care visits over a period of 5 years post-implantation. All assessments of the registry are part of the standard clinical care. Data collection will include polysomnographic data, home sleep test data, therapy usage, device data and questionnaires (Epworth Sleepiness Scale, Functional Outcomes of Sleep Questionnaire-30, Visual Analogue Scale (VAS) snoring.

Data will be collected from routine visits including: pre-implant, implant, activation, titration, follow-up (6, 12, 24, 36, 48 and 60 months post-implantation).

ELIGIBILITY:
Inclusion Criteria:

Any patient implanted with or receiving the Inspire HNS system and who is able to give informed consent is eligible to participate in the registry. A patient is eligible for HNS implantation if he/she meets the following criteria:

* At least 18 years old at the time of implantation
* The patient suffers from moderate to severe OSA (15 events/h ≤ AHI ≤ 65 events/h)
* The patient has failed, not tolerated or has a contraindication for continuous positive airway pressure (CPAP) and/or mandibular advancement device (MAD) therapy
* Absence of complete concentric collapse of the level of the soft palate during Drug-Induced Sleep Endoscopy (DISE)

Exclusion Criteria:

* Body mass index (BMI) >32 kg/m².
* Combined mixed and central AHI is more than 25% of the total AHI
* Patients with complete concentric collapse at the level of the soft palate or any other anatomical deviation that could impede the proper functioning of HNS
* Patients with severely impaired neurological control over the upper airway
* Pregnancy
* Surgery performed on the soft palate in the past three months before implantation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient implanted with or receiving HNS therapy in routine clinical care in Belgium and that is able to give informed consent is eligible to participate in the registry.
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2034-04 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Delta apnea-hypopnea index (AHI) as measured by a polysomnography | From baseline to 6, 12 and 60 months post-implantation
  The AHI is an index of sleep apnea severity that encompasses the frequency of apneas (cessations in breathing) and hypopneas (reductions in airflow) per hour of sleep.

SECONDARY OUTCOMES:
% of patients that reach treatment success defined by a 50% reduction in AHI and an on therapy AHI of < 20 events/h OR an on therapy AHI of < 15 events/h | At 6, 12 and 60 months post-implantation
  AHI is determined during a polysomnography
Therapy adherence defined by the amount of hours therapy usage per night. | At 6, 12 and 60 months post-implantation
  Average hours of therapy use per night can be retrieved from data stored in the device
Delta oxygen desaturation index (ODI) as measured by a polysomnography | From baseline to 6, 12 and 60 months post-implantation
  The ODI represents the average number of desaturation episodes (≥3%) per hour sleep and will be determined during a polysomnography.
Daytime sleepiness measured by the Epworth Sleepiness Scale (ESS) questionnaire | From baseline to 6, 12 and 60 months post-implantation
  The ESS questionnaire assesses the probability of falling asleep in various settings and situations in daily life. This questionnaire consists of eight questions which can be scored on a four-point Likert-type scale. The lowest score (zero) suggests that the described incident is absent and the highest score (three) suggests the presence of this event. The summation of the eight items can range from 0 to 24.
Disease-specific quality of life as measured by the Functional Outcomes of Sleep Questionnaire-30 (FOSQ-30) questionnaire | From baseline to 6, 12 and 60 months post-implantation
  The FOSQ-30 is a disease-specific quality of life questionnaire that determines functional status in adults; measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living and the extent to which these abilities are improved by effective treatment.
Degree of snoring measured by the Visual Analogue Scale (VAS) questionnaire | From baseline to 6, 12 and 60 months post-implantation
  Snoring intensity is evaluated using a 10 cm visual analogue scale (VAS) from 0 to 10: 0 represents no snoring, 1-3 represents minimally annoying, 4-6 represents moderately annoying, 7-9 represents annoying, and 10 represents extremely annoying
Flow-derived site of collapse | At 6, 12 and 60 months post-implantation
  Several parameters extracted from the flow signal, including negative effort dependence (NED), peak inspiratory flow, etc. measured during routine polysomnography
Pathophysiological endotypes | At 6, 12 and 60 months post-implantation
  Changes in pathophysiological traits (Vpassive, Vactive, Arousal Threshold, Loop Gain) will be quantified as %Veupnea from polysomnography data using a validated algorithm.
New OSA severity metrics | At 6, 12 and 60 months post-implantation
  Change in sleep apnea specific hypoxic burden (SASHB), delta heart rate and pulse wave amplitude drops.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Vanderveken, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (2):
- Belgium (2):
  - Antwerp University Hospital, Edegem, Antwerp
  - AZ Sint-Jan Brugge, Bruges, West-Vlaanderen